CLINICAL TRIAL: NCT01007500
Title: Effect of Dexamethasone Combined With Ondansetron on Postoperative Nausea and Vomiting in Patients With Patient-controlled Analgesia After Video-assisted Thoracoscopic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Shim, Yon Hee/associate professor, Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Reseach Institute, Yonsei University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2009-0407
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Nausea; Vomiting
Keywords: Postoperative nausea and vomiting after video-assisted thoracoscopic surgery
MeSH Terms: conditions — Nausea; Vomiting; Postoperative Nausea and Vomiting | interventions — Dexamethasone; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone
- Group Ondansetron (Active Comparator)
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Dexamethasone — Experimental: Dexamethasone 8 mg IV after induction of anesthesia, Ondansetron 4 mg IV at the end of surgery and 12 mg mix to intravenous patient controlled analgesia device.
  Arms: Group Dexamethasone
Drug: Ondansetron — Active comparator: Ondansetron 4 mg IV at the end of surgery and 12 mg mix to intravenous patient controlled analgesia device.
  Arms: Group Ondansetron

SUMMARY:
The purpose of this study is to study the effect of dexamethasone combined with ondansetron on postoperative nausea and vomiting in patients with patient-controlled analgesia after video-assisted thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing video-assisted thoracoscopic surgery
* Age 20-75
* American Society of Anesthesiologists physical status classification I or II

Exclusion Criteria:

* Antiemetic within 24 hrs
* Taking Steroids, Opioids within 1 week
* Active drug or alcohol abuse
* GI motility disorder, severe renal/ hepatic disease.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | within 48 hrs after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea